CLINICAL TRIAL: NCT02749253
Title: Sudarshan Kriya Yoga (SKY) in Post Traumatic Stress Disorder: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Kamini Vasudev, Dr. Kamini Vasudev, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107728
Record Dates: First submitted 2016-03-06; First posted 2016-04-22 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder (PTSD); Sudarshan Kriya Yoga (SKY)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sudarshan Kriya Yoga Trauma Relief Program (SKY) (Experimental): Participants will receive training in SKY soon after completing baseline assessments.
  Interventions: Other: Sudarshan Kriya Yoga Tauma Relief Program (SKY).

INTERVENTIONS:
Other: Sudarshan Kriya Yoga Tauma Relief Program (SKY). — Sudarshan Kriya Yoga Trauma Relief Program (SKY) participants will undergo a 12-week training course in SKY conducted by certified instructors from the Art of Living Foundation

SUMMARY:
This pilot study is designed to investigate the feasibility of sudarshan kriya yoga (SKY) program in adults with post traumatic stress disorder (PTSD) resulting from a wide range of trauma experience.

SKY incorporates standardized collection of breathing techniques which are known to positively influence the autonomic nervous system and stress response system. Both these systems are dysregulated in PTSD.

DETAILED DESCRIPTION:
This is a single-center, open-label,longitudinal, empirical, feasibility trial of a 12 week intervention of Sudarshan Kriya Yoga in patients with Post traumatic stress disorder.

Research participants will be men and women, 18-75 years of age, who have a confirmed diagnosis of PTSD. Recruitment will occur from the general adult ambulatory mental health clinics as well as the geriatric mental health program in London.

Potential participants will be screened as per inclusion and exclusion criteria by trained research staff. These patients will already have a clinically diagnosed PTSD by a psychiatrist and any other co-morbid diagnoses would have been previously confirmed by the physician. However, for research purposes a diagnosis of PTSD will be confirmed through a structured clinical interview specifically the MINI (Mini International neuropsychiatric Interview) and the Clinician-administered PTSD Scale for DSM5- past month version (CAPS5). CAPS5 will also be used to rule out exclusion criteria of severe depersonalization and derealization. The scales will be administered by a trained research staff and confirmed by a psychiatrist. The MINI will also be used to assess for presence of current suicidality. If the total score on Questions C1 and C2 is more than 5 then this will be reported to the PI who will further assess the patient for safety and risk assessment. If the participant is above the age of 65 years of age they will also be asked to complete a cognitive screening test (Mini Mental State Examination, MMSE) to ensure they are not suffering from any significant cognitive impairment

A 12-week intervention of Sudarshan Kriya Yoga will be conducted, as per the details provided below. The SKY PTSD program is a mind-body resilience building program which has been specifically developed for persons with PTSD by the investigators collaborating not for profit organisation, Art of Living Foundation. The investigators wish to assess the feasibility of this intervention in the investigators routine trauma clinic at LHSC. The prescribed program of SKY includes specific breathing exercises, interactive discussions, journaling, yoga and guided meditations. It is supposed that the workshop builds a framework for resilience and empowerment, and develops self-awareness, connectedness and community, and a positive outlook. This minimally invasive treatment is not routinely performed as part of standard of care and is being applied in the study population for research purposes only. In addition to using feasibility measures, the investigators will use well-established clinical scales to assess symptoms of PSTD as well as comorbid depression, anxiety, quality of life as well as physiological measurements of the heart. These specifically include heart rate variability (HRV) and blood pressure measured at baseline (week 0), week 12 and week 24. Additionally, the investigators shall collect blood samples to measure possible changes in blood inflammatory markers at these three intervals of the study as described below.

Sudarshan Kriya Yoga (SKY): Participants will continue to receive their treatment as usual, including pharmacotherapy and/or psychotherapy. Following the initial clinical screening measurements, participants will undergo a 12-week training course conducted by certified instructors from the Art of Living Foundation who will be supervised by one of the study co-investigators (RN). There will be two instructors for this study (one male Spenser Delisle and one female Hiteshini Jugessur) for the initial 6 day course; both are certified as Art of Living instructors of SKY, in addition to being certified to work with traumatized populations. They have had experience of teaching more than 2000 people in multiple settings. Additional certified instructors may conduct follow up sessions. There will always be an overlap between the existing instructor and a replacement instructor, to ensure comfort of study participants. SKY training will take place in group-format (group sizes of 8-15 participants) in an appropriately sized and accessible community hall in London, Ontario. Given that men and women tend to have different sources of trauma, separate groups will be held for each gender. This is in accordance with current practices used in the Trauma Program at LHSC. While the investigators do not anticipate gender differences, the investigators have decided to stratify this study by gender to allow participants in these groups to feel more safe and comfortable, which is key to maximizing benefits of the course. SKY training involves attending a week-long (6 days) course that teaches the basic principles of SKY over 2.5-3 hour daily sessions. This will be followed by once weekly follow up sessions (90 min/wk) for 3 weeks and then bimonthly sessions (every 2 weeks) for the next 8 weeks. In addition, participants will be asked to practice SKY at home daily (25 min/day) throughout the duration of the study period and log practice frequency and any other noteworthy observations in a log sheet that will be provided to them (please see attached log sheet). Nutritional snacks will be provided during the 6 session SKY training course. Information regarding demographic data, past psychiatric history, current ongoing psychological interventions, current medications, smoking and substance use status and any comorbid medical illnesses will be collected at baseline. Any change in status of ongoing psychological interventions, medications, smoking, alcohol and substance use, medical illnesses will be noted at each assessment visit in addition to hospitalizations or ER visits. This information is important to control for confounding factors as well as for risk assessment. The weight and height of patients will be measured at baseline and weight will be measured at each assessment visit to monitor for any effect of SKY yoga on weight (positive or negative). The information will be asked from the patient and/ or collected from the clinical charts if patient is distressed about giving the information, particularly past psychiatric history including trauma. Any adverse effects related to SKY will be monitored using a structured questionnaire, at each assessment visit (week 4, 8, 12 and 24).

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of PTSD as per CAPS5 (Clinician Administered PTSD Scale for DSM 5- past month version) criteria.
2. If participants are using antidepressants or antipsychotics used as mood augmenting agents, they must be at therapeutic doses for a minimum of four weeks prior to commencing the study. Patients who are not willing to take any medications will also be eligible for the study
3. Sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 60 minutes.
4. Willing and able to attend 6 initial SKY training sessions and 75% of follow up sessions
5. Not pregnant and willing to remain not pregnant for the duration of the study

Exclusion Criteria:

1. They are currently participating in a similar study on either a pharmacological or non-pharmacological intervention for treatment of their PTSD.
2. If the patient scores severe or extreme on Depersonalization (item 29) or Derealization (item 30) items of CAPS5.
3. Other significant mental health diagnosis including substance dependence, Major Neurocognitive disorder, Panic Disorder, Bipolar disorder and/or Personality disorder (confirmed by Psychiatrist and MINI)
4. High risk of suicide as elicited by clinical interview (MINI).
5. Psychotic episodes within the past 12 months.
6. Traumatic Brain Injury (TBI) as defined by loss of consciousness for more than 20 minutes and/or Glasgow Coma Scale score less than or equal to 12. The researcher will use self-reported histories to screen for traumatic brain injury and if necessary confirmed by medical records.
7. Currently practicing any type of formal meditation, mindfulness or breathing techniques regularly.
8. Serious cardiovascular disease in the past 12 months (i.e. myocardial infarction, stroke, TIA, uncontrolled hypertension), or a past history of neurological disease (including Parkinson's Disease), seizures, or diabetic neuropathy
9. Major surgery within 6 weeks prior to commencement of the intervention, or a scheduled major surgery during the intervention period. (This is due to the physical rigor of the breathing techniques)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the number of potential participants approached. | 2 years
  The number of potential participants with PTSD who are approached for potential study participation will be recorded. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the proportion of participants successfully screened. | 2 years
  The proportion of successfully screened participants with PTSD will be recorded. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the proportion of screened participants who enroll. | 2 years
  The proportion of screened participants with PTSD who enroll will be recorded. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the retention rate of the study. | 2 years
  The proportion of participants enrolled in the study who complete the study intervention and assessments will be assessed. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the rate of adherence to study protocol. | 2 years
  Participant intervention attendance and assessment attendance will be recorded to determine if participants are willing to adhere to the study protocol. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the proportion of completed planned ratings. | 2 years
  The proportion of completed planned ratings will be calculated. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the intervention cost per case. | 2 years
  The intervention cost per study participant will be calculated. This information will be used to assess if a larger SKY study for participants with PTSD is financially feasible.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the completeness of final data for analysis. | 2 years
  The completeness of final data for analysis will be assessed. The proportion of incomplete Case Report Forms and Questionnaires will be calculated. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for Sudarshan Kriya Yoga Trauma Relief Program (SKY) in participants with Post Traumatic Stress Disorder (PTSD) considering the length of time to collect all data. | 2 years
  The length of time to collect all data will be recorded, including the time required for each assessment, and the time required to enter data into a database. The proportion of incomplete Case Report Forms and Questionnaires will be calculated. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for SKY in participants with PTSD considering any capacity issues with partners providing intervention and investigators being able to perform the tasks that they are committed to doing. | 2 years
  Any capacity issues with the partners providing intervention and investigators being able to perform the tasks that they are committed to doing will be recorded. This information will be used to assess if a larger SKY study for participants with PTSD is likely to be successful.
Feasibility of conducting a larger RCT for SKY in participants with Post Traumatic Stress Disorder (PTSD) considering if it is safe to apply the intervention in this population as assessed by a SKY adverse effects questionnaire. | 2 years
  A SKY adverse effects questionnaire will be used at baseline, week 4, week 8, and week 12 to assess if the SKY intervention is safe to use in this population. This information will be assessed at two years and used to determine if a larger SKY study for participants with PTSD is likely to be successful.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No